CLINICAL TRIAL: NCT03356665
Title: Diagnostic Tools for Human African Trypanosomiasis Elimination and Clinical Trials: WP2 Passive Case Detection
Acronym: DiTECT-WP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Ministry of Public Health, Democratic Republic of the Congo (Other Government); Ministry of Health, Guinea (Other Government); Institut National de Sante Publique (Other); Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); CIRDES (Unknown); Institute of Tropical Medicine, Belgium (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DiTECT-HAT-WP2
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: African Trypanosomiases; West African; Trypanosomiasis; Sleeping Sickness; West African; Trypanosoma Brucei Gambiense; Infection
Keywords: diagnosis; sensitivity; specificity; rapid diagnostic test; molecular biology; LAMP; RT-PCR; serology; ELISA; immune trypanolysis; clinical symptom
MeSH Terms: conditions — Trypanosomiasis, African; Trypanosomiasis; Infections; Disease; Hypersensitivity | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Intervention Model Description: Sequential assignement
Masking Description: The reference laboratory, generating the results for 4 index tests, is masked for index test and reference test results obtained at the clinical trial site
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical suspect (Experimental): Diagnostic tests: Rapid diagnostic test (RDT); Serological and molecular tests on DBS
  Interventions: Diagnostic Test: Rapid diagnostic test (RDT); Diagnostic Test: Serological and molecular tests on DBS

INTERVENTIONS:
Diagnostic Test: Rapid diagnostic test (RDT) — The 4 rapid diagnostic tests (RDT) will be carried out on fresh blood from clinical suspects. Only those subjects that are positive in at least 1 RDT will 1) undergo tests on DBS (immune trypanolysis, ELISA and DNA detection); 2) undergo parasitological confirmation (reference standard) at inclusion.
  Other Names: rHAT Sero-Strip (Coris Bioconcept, Belgium); SD Bioline HAT 1.0 (Standard Diagnostics Korea); HAT Sero-K-Set (Coris Bioconcept, Belgium); SD Bioline HAT 2.0 (Standard Diagnostics Korea)
Diagnostic Test: Serological and molecular tests on DBS — Serological and molecular reference tests on dried blood spots (DBS) are carried out on RDT positive clinical suspects, which also undergo parasitological examination at inclusion (reference standard). If at least one of the serological or molecular reference tests on dried blood spots is positive, parasitological examination is repeated 3 and 6 months after inclusion. The combined results of parasitological examinations (at inclusion and if applicable at 3 and 6 months) serve as reference standard
  Other Names: Immune trypanolysis: presence of antibodies; ELISA: on native LiTat 1.3 + LiTat 1.5 VSG; Loopamp T. brucei Detection Kit (Eiken); RT-PCR: Trypanozoon 18S, Tbg TgsGP

SUMMARY:
The study determines the diagnostic performance and cost of rapid diagnostic tests (RDTs) performed on human African trypanosomiasis clinical suspects in peripheral health centres, whether or not followed by serological and/or molecular tests on dried blood spots done at regional reference centres

DETAILED DESCRIPTION:
In the last decade, the prevalence of Trypanosoma brucei gambiense human African trypanosomiasis (HAT) has fallen and HAT has been targeted for elimination. At low disease prevalence, integration of case finding into routine activities of peripheral health centres becomes crucial. However, HAT case detection by the peripheral health system with limited resources requires adapted diagnostic tests and test algorithms.

The objective of the DiTECT-HAT-WP2 study is to determine the diagnostic performance and cost of rapid diagnostic tests (RDTs) performed on clinical suspects in peripheral health centres, whether or not followed by serological and/or molecular tests on filter paper done at regional reference centres.

The DiTECT-HAT-WP2 study will be conducted in centres for diagnosis and treatment and in sites for serological screening in Guinea, Côte d'Ivoire and DR Congo. In these centres and sites, clinical suspects will be tested with several commercially available RDTs for HAT. Clinical suspects with at least 1 RDT positive result, will 1° undergo parasitological examination and 2° blood collection on filter paper for reference analysis in trypanolysis, LAMP, ELISA and real-time PCR in the regional reference laboratory. If the reference laboratory tests and parasitological examinations are all negative, the suspect is informed and considered free of HAT. If at least 1 reference test is positive, parasitological examinations are repeated at least twice at three months interval, unless trypanosomes are detected. In order to assess the sensitivity, specificity, Positive Predictive Values and Negative Predictive Values of each assay in these multiple populations, the data from the multiple assays in the 3 countries will be used in a Bayesian formulation of the Hui-Walter latent class model, to estimate the assay performances in the absence of a gold standard. As we will collect full cost information for the different algorithms, we will, in addition to estimating the diagnostic effectiveness of the assay, be able to estimate the cost of each assay in each setting, and rank this jointly with assay performance.

The results will enable us to propose cost-effective test algorithms to detect HAT, adapted to peripheral health centres. Algorithms with high positive predictive values might allow test-and-treat scenarios without the need for complicated parasitological confirmations, once safe oral easy to use drugs become available to treat HAT.

ELIGIBILITY:
Inclusion Criteria:

* Visit of or residence in a HAT endemic area
* Clinical suspicion of HAT based on: Recurrent fever not responding to anti-malarial medication; or Headache for a long duration (>14 days); or presence of swollen lymph nodes in the neck; or Important weight loss; or Weakness; or Important scratching; or Amenorrhea, abortion(s), or sterility; or Coma; or Psychiatric problems (aggressiveness, apathy, mental confusion, increasing unusual hilarity, ...); or Sleep disruption (nocturnal insomnia and excessive diurnal sleeping); or Motor abnormalities (convulsions, abnormal movements, shaking, walking difficulties); or Speech disorders.

Exclusion Criteria:

* Previously treated for HAT (irrespective of time elapsed since treatment)
* No informed consent
* < 4 years old

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10700 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity for HAT diagnosis of RDT, RDT combinations, algorithms of RDT and serological and/or molecular tests on HAT clinical suspects | 6 months
  Index tests: 4 RDTs on fresh blood, and for RDT positives also immune trypanolysis on DBS, ELISA on DBS, LAMP on DBS, RT-PCR on DBS.
  Reference standard: for RDT positives only: combined results of parasitological examination at inclusion and if one of tests on DBS positive, at 3 and 6 months. Subjects negative in all RDTs are considered HAT negative
Specificity for HAT diagnosis of RDT, RDT combinations, algorithms of RDT and serological and/or molecular tests on HAT clinical suspects | 6 months
  Index tests: 4 RDTs on fresh blood, and for RDT positives also immune trypanolysis on DBS, ELISA on DBS, LAMP on DBS, RT-PCR on DBS.
  Reference standard: for RDT positives only: combined results of parasitological examination at inclusion and if one of tests on DBS positive, at 3 and 6 months. Subjects negative in all RDTs are considered HAT negative.

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Lejon, PhD, Principal Investigator — Institut de Recherche pour le Developpement
Locations (3):
- Institut Pierre Richet, Institut National de Santé Publique, Bouaké, Côte d’Ivoire
- Programme Nationale de Lutte contre la trypanosomiase humaine Africaine, Kinshasa, Democratic Republic of the Congo
- Programme Nationale de Lutte contre la Trypanosomiase Humaine Africaine, Ministère de Santé, Division Prévention et Lutte contre la Maladie, Conakry, Guinea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bisser S, Lumbala C, Nguertoum E, Kande V, Flevaud L, Vatunga G, Boelaert M, Buscher P, Josenando T, Bessell PR, Bieler S, Ndung'u JM. Sensitivity and Specificity of a Prototype Rapid Diagnostic Test for the Detection of Trypanosoma brucei gambiense Infection: A Multi-centric Prospective Study. PLoS Negl Trop Dis. 2016 Apr 8;10(4):e0004608. doi: 10.1371/journal.pntd.0004608. eCollection 2016 Apr. PMID 27058033
- [Background] Buscher P, Deborggraeve S. How can molecular diagnostics contribute to the elimination of human African trypanosomiasis? Expert Rev Mol Diagn. 2015 May;15(5):607-15. doi: 10.1586/14737159.2015.1027195. Epub 2015 Mar 18. PMID 25786994
- [Background] Buscher P, Mertens P, Leclipteux T, Gilleman Q, Jacquet D, Mumba-Ngoyi D, Pyana PP, Boelaert M, Lejon V. Sensitivity and specificity of HAT Sero-K-SeT, a rapid diagnostic test for serodiagnosis of sleeping sickness caused by Trypanosoma brucei gambiense: a case-control study. Lancet Glob Health. 2014 Jun;2(6):e359-63. doi: 10.1016/S2214-109X(14)70203-7. Epub 2014 May 9. PMID 25103304
- [Background] Camara O, Camara M, Lejon V, Ilboudo H, Sakande H, Leno M, Buscher P, Bucheton B, Jamonneau V. Immune trypanolysis test with blood spotted on filter paper for epidemiological surveillance of sleeping sickness. Trop Med Int Health. 2014 Jul;19(7):828-31. doi: 10.1111/tmi.12316. Epub 2014 Apr 18. PMID 24750463
- [Background] Hasker E, Lutumba P, Mumba D, Lejon V, Buscher P, Kande V, Muyembe JJ, Menten J, Robays J, Boelaert M. Diagnostic accuracy and feasibility of serological tests on filter paper samples for outbreak detection of T.b. gambiense human African trypanosomiasis. Am J Trop Med Hyg. 2010 Aug;83(2):374-9. doi: 10.4269/ajtmh.2010.09-0735. PMID 20682885
- [Background] Jamonneau V, Bucheton B, Kabore J, Ilboudo H, Camara O, Courtin F, Solano P, Kaba D, Kambire R, Lingue K, Camara M, Baelmans R, Lejon V, Buscher P. Revisiting the immune trypanolysis test to optimise epidemiological surveillance and control of sleeping sickness in West Africa. PLoS Negl Trop Dis. 2010 Dec 21;4(12):e917. doi: 10.1371/journal.pntd.0000917. PMID 21200417
- [Background] Jamonneau V, Camara O, Ilboudo H, Peylhard M, Koffi M, Sakande H, N'Dri L, Sanou D, Dama E, Camara M, Lejon V. Accuracy of individual rapid tests for serodiagnosis of gambiense sleeping sickness in West Africa. PLoS Negl Trop Dis. 2015 Feb 2;9(2):e0003480. doi: 10.1371/journal.pntd.0003480. eCollection 2015 Feb. PMID 25642701
- [Background] Mitashi P, Hasker E, Mbo F, Van Geertruyden JP, Kaswa M, Lumbala C, Boelaert M, Lutumba P. Integration of diagnosis and treatment of sleeping sickness in primary healthcare facilities in the Democratic Republic of the Congo. Trop Med Int Health. 2015 Jan;20(1):98-105. doi: 10.1111/tmi.12404. Epub 2014 Oct 20. PMID 25329353
- [Background] Mitashi P, Hasker E, Ngoyi DM, Pyana PP, Lejon V, Van der Veken W, Lutumba P, Buscher P, Boelaert M, Deborggraeve S. Diagnostic accuracy of loopamp Trypanosoma brucei detection kit for diagnosis of human African trypanosomiasis in clinical samples. PLoS Negl Trop Dis. 2013 Oct 17;7(10):e2504. doi: 10.1371/journal.pntd.0002504. eCollection 2013. PMID 24147176
- [Background] Mumba D, Bohorquez E, Messina J, Kande V, Taylor SM, Tshefu AK, Muwonga J, Kashamuka MM, Emch M, Tidwell R, Buscher P, Meshnick SR. Prevalence of human African trypanosomiasis in the Democratic Republic of the Congo. PLoS Negl Trop Dis. 2011 Aug;5(8):e1246. doi: 10.1371/journal.pntd.0001246. Epub 2011 Aug 2. PMID 21829736
- [Background] Njiru ZK. Loop-mediated isothermal amplification technology: towards point of care diagnostics. PLoS Negl Trop Dis. 2012;6(6):e1572. doi: 10.1371/journal.pntd.0001572. Epub 2012 Jun 26. No abstract available. PMID 22745836
- [Background] Van Meirvenne N, Magnus E, Buscher P. Evaluation of variant specific trypanolysis tests for serodiagnosis of human infections with Trypanosoma brucei gambiense. Acta Trop. 1995 Dec;60(3):189-99. doi: 10.1016/0001-706x(95)00127-z. PMID 8907397
- [Derived] Makabuza J, Lukusa IN, Lumbala C, Miaka EM, Nganzobo P, Fukinsia A, Kwete J, Bebronne N, Buscher P, Ngoyi DM, Lejon V. Passive surveillance of human African trypanosomiasis in the Democratic Republic of the Congo: clinical presentation and prospective evaluation of rapid diagnostic and reference laboratory test accuracy. PLoS Negl Trop Dis. 2025 Sep 29;19(9):e0013045. doi: 10.1371/journal.pntd.0013045. eCollection 2025 Sep. PMID 41021650
- [Derived] Camara O, Camara M, Falzon LC, Ilboudo H, Kabore J, Compaore CFA, Fevre EM, Buscher P, Bucheton B, Lejon V. Performance of clinical signs and symptoms, rapid and reference laboratory diagnostic tests for diagnosis of human African trypanosomiasis by passive screening in Guinea: a prospective diagnostic accuracy study. Infect Dis Poverty. 2023 Mar 20;12(1):22. doi: 10.1186/s40249-023-01076-1. PMID 36941656
- [Derived] Kone M, Kaba D, Kabore J, Thomas LF, Falzon LC, Koffi M, Kouame CM, Ahouty B, Compaore CFA, N'Gouan EK, Solano P, Fevre E, Buscher P, Lejon V, Jamonneau V. Passive surveillance of human African trypanosomiasis in Cote d'Ivoire: Understanding prevalence, clinical symptoms and signs, and diagnostic test characteristics. PLoS Negl Trop Dis. 2021 Aug 30;15(8):e0009656. doi: 10.1371/journal.pntd.0009656. eCollection 2021 Aug. PMID 34460829